CLINICAL TRIAL: NCT01704417
Title: A Trial Comparing the Effect of Exercise on Blood Glucose Between Insulin Degludec and Insulin Glargine in Subjects With Type 1 Diabetes
Brief Title: A Trial Comparing the Effect of Exercise on Blood Glucose in Subjects With Type 1 Diabetes, Who Are Treated With Either Insulin Degludec or Insulin Glargine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3999; 2012-000329-37 (EudraCT Number); U1111-1127-3402 (Other: WHO)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg followed by IGlar (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine
- IGlar followed by IDeg (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Subjects will be randomised to a treatment sequence consisting of two treatment periods in which the subjects will receive IDeg and IGlar, respectively. Administered subcutaneously (s.c., under the skin) once daily. Dose individually adjusted.
Drug: insulin glargine — Subjects will be randomised to a treatment sequence consisting of two treatment periods in which the subjects will receive IDeg and IGlar, respectively. Administered subcutaneously (s.c., under the skin) once daily. Dose individually adjusted.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to compare the effect of exercise on blood glucose in subjects with type 1 diabetes, who are treated with either insulin degludec (IDeg) or insulin glargine (IGlar).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-27.0 kg/m^2 (both inclusive)
* Subjects performing regular physical cardiorespiratory activity
* Glycosylated haemoglobin (HbA1c) below or equal to 9.5 %

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period
* Supine blood pressure at screening (after resting for at least 5 minutes) outside the range of 90-140 mmHg for systolic or 50-90 mmHg for diastolic

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
BGpre-exe - BGminimum,exe, difference between blood glucose concentration before exercise and the minimum blood glucose concentration observed during exercise | From 0 to 30 minutes

SECONDARY OUTCOMES:
BGmean,exe, mean blood glucose concentration during exercise | From 0 to 30 minutes
BGmean,30-180min,post-exe, mean blood glucose concentration | Between 30 and 180 minutes, i.e. post-exercise
BGminimum,30-180min,post-exe, minimum blood glucose concentration | Between 30 and 180 minutes, i.e. post-exercise

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Bain SC, Bracken RM, Zijlstra E, Nosek L, Stender-Petersen K, Rabol R, Rowe E, Haahr HL. Similar risk of exercise-related hypoglycaemia for insulin degludec to that for insulin glargine in patients with type 1 diabetes: a randomized cross-over trial. Diabetes Obes Metab. 2016 Feb;18(2):196-9. doi: 10.1111/dom.12588. Epub 2015 Nov 27. PMID 26450456
- [Derived] McCarthy O, Pitt J, Wellman B, Eckstein ML, Moser O, Bain SC, Bracken RM. Blood Glucose Responses during Cardiopulmonary Incremental Exercise Testing in Type 1 Diabetes: A Pooled Analysis. Med Sci Sports Exerc. 2021 Jun 1;53(6):1142-1150. doi: 10.1249/MSS.0000000000002584. PMID 33315813
- [Derived] Eckstein ML, Farinha JB, McCarthy O, West DJ, Yardley JE, Bally L, Zueger T, Stettler C, Boff W, Reischak-Oliveira A, Riddell MC, Zaharieva DP, Pieber TR, Muller A, Birnbaumer P, Aziz F, Brugnara L, Haahr H, Zijlstra E, Heise T, Sourij H, Roden M, Hofmann P, Bracken RM, Pesta D, Moser O. Differences in Physiological Responses to Cardiopulmonary Exercise Testing in Adults With and Without Type 1 Diabetes: A Pooled Analysis. Diabetes Care. 2021 Jan;44(1):240-247. doi: 10.2337/dc20-1496. Epub 2020 Nov 12. PMID 33184152
- [Derived] Moser O, Eckstein ML, McCarthy O, Deere R, Bain SC, Haahr HL, Zijlstra E, Bracken RM. Poor glycaemic control is associated with reduced exercise performance and oxygen economy during cardio-pulmonary exercise testing in people with type 1 diabetes. Diabetol Metab Syndr. 2017 Nov 21;9:93. doi: 10.1186/s13098-017-0294-1. eCollection 2017. PMID 29201153
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com